CLINICAL TRIAL: NCT01217515
Title: A Randomised,Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of Diltiazem Hydrochloride Cream in Subjects With Anal Fissure
Brief Title: Diltiazem Hydrochloride Cream for Anal Fissure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: S.L.A. Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-AF-09
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Anal Fissure
MeSH Terms: interventions — Diltiazem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diltiazem hydrochloride 4% cream (Experimental): 2.5 cm Diltiazem hydrochloride 4% cream applied peri-anally three times daily for eight weeks.
  Interventions: Drug: Diltiazem hydrochloride 4% cream
- Diltiazem hydrochloride 2% cream (Experimental): 2.5 cm of Diltiazem hydrochloride 2% cream applied peri-anally three times daily for eight weeks.
  Interventions: Drug: Diltiazem hydrochloride 2% cream
- Placebo cream (Placebo Comparator): 2.5 cm placebo cream applied peri-anally three times daily for eight weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Diltiazem hydrochloride 4% cream — 3 times daily
  Arms: Diltiazem hydrochloride 4% cream
Drug: Diltiazem hydrochloride 2% cream — 3 times daily
  Arms: Diltiazem hydrochloride 2% cream
Other: Placebo — 3 times daily
  Arms: Placebo cream

SUMMARY:
A Phase III, multicentre, randomised, double blind, placebo-controlled study in subjects having anal fissure (AF) with AF-related pain. Subjects will undertake a 1-week screening period to provide baseline data and for assessment of eligibility. At the Baseline visit (Week 0), eligible subjects (having an average Numerical Rating Scale (NRS) score of >4 for worst pain associated with or following defaecation) will be randomised on a 1:1:1 basis to one of the three treatment groups. Subjects will receive diltiazem hydrochloride 2% cream or diltiazem hydrochloride 4% cream or placebo cream. Study treatment will be applied in and around the anus, three times daily, for up to 8 weeks. Following the Week 0 Visit, subjects will be contacted by telephone during Week 1 to ensure adequate compliance with study treatment, to ensure that study drug is being tolerated and that any concomitant medications are used at a level consistent with that prior to randomisation. Subjects will return to the clinic for safety and efficacy assessments at Weeks 2, 4, and 8 and receive a follow-up telephone call at Week 12, following cessation of therapy.

Concomitant laxatives and stool softeners will be permitted, as needed, during the entire study period (screening and treatment) to ensure that constipation or passage of hard stools does not confound evaluation or improvement of the condition. Fibre supplements will be allowed but should be continued at the baseline level.

Instructions on the use of the Interactive Voice Response System (IVRS) diary will be issued to subjects to record fissure-related pain (NRS) and bowel symptoms daily during the 1-week screening period, to confirm eligibility and post-randomisation to record worst anal pain associated with or following defaecation (NRS) and daily overall AF-related pain (NRS). A record of the number of times the subject has defaecated, laxative and analgesic usage will also be made as well as the number of applications of study treatment, any changes to concurrent medications and any Adverse Events (AEs).

In addition, at some or all study visits, subjects will record the Patient's Global Impression of Improvement (PGI-I) on a 7 point Likert scale, complete a Short Form 36 (SF-36) quality of life questionnaire and will undergo examination of their AF. Routine blood samples will be taken and the Skin Irritation Score (SIS) recorded for safety evaluations.

Subjects may receive permitted medications for pain per Entry Criteria, but these should remain stable, where possible, up to the Week 8 Visit. Introduction of any new medication for AF will not be permitted unless the Investigator deems "rescue" intervention necessary. A subject will be deemed a treatment failure if rescue intervention is required and will have to be withdrawn from the study.

Any subject leaving the study following randomisation for any reason will be asked to complete the Early Withdrawal Visit. This includes subjects who withdraw due to the development of AEs or intolerance, as well as subjects who require rescue intervention. These subjects will return for safety follow-up visits at their previously scheduled follow-up assessment appointments. If complete healing has occurred at the 2 or 4 Week visits, (i.e. prior to the end of the 8-week treatment period), subjects will be asked to continue applying the medication for the full 8 week course, up to the final assessment.

Following the Week 8 visit (or Early Withdrawal Visit), subjects will be followed up for a further 4 weeks (following cessation of study medication) to note any AEs.

All routine blood analyses (haematology and biochemistry) and plasma levels of diltiazem and of its principal metabolites will be analysed by central laboratories.

ELIGIBILITY:
Inclusion Criteria:

* • Must give written informed consent.

  * Male or female subjects, from 18 years of age.
  * Subjects with at least a 4 week history of painful AF, prior to screening, where AF-related pain associated with, or following, defaecation is experienced at least twice a week for the 4 weeks prior to Screening with an average of ≥ 3 on an 11-point NRS (Numerical Rating Scale, range 0-10 where 0 = no pain and 10 = worst pain imaginable).
  * Subjects with an average of ≥4 on an 11-point NRS during the screening phase for worst anal pain associated with, or following, defaecation for the most recent 3 days on which the subject has defaecated.
  * Subjects with evidence of a circumscribed fissure, with induration at the edges.
  * Willing to stop all other concomitant topical preparations applied perianally prior to commencing study treatment, and throughout the study.
  * Willingness and ability to use the IVRS diary.

Exclusion Criteria:

* Subjects unwilling to have examination of AF.
* Subjects with "acute" AF (i.e. duration of symptoms less than 4 weeks prior to screening, and/or no induration of fissure edges).
* More than 1 AF.
* Subjects who have had lateral sphincterotomy or anal stretch or other previous surgery involving the anal canal or perianal region.
* Subjects who have had sub-fissure injection of botulinum toxin in the 3 months prior to screening, or have used glyceryl trinitrate (GTN) ointment for >1 week in the 4 weeks prior to the screening visit.
* Subjects with AF associated with other conditions (drug-induced [e.g. nicorandil], trauma, HIV infection, fistula-in-ano, inflammatory bowel disease, perianal sepsis or malignancy).
* Subjects with cardiovascular disease (including those diagnosed by the screening ECG): history of reduced left ventricular function, bradycardia, 1st degree atrioventricular (AV) block or prolonged P-R interval (>0.2 seconds/ >200 milliseconds).
* Subjects with known hypersensitivity to diltiazem.
* Subjects who have previously received therapy with diltiazem hydrochloride cream or other topical calcium channel blockers.
* Subjects taking medications prohibited by the protocol.
* Subjects who have taken experimental agents must have been discontinued at least 8 weeks prior to screening, or for a period equivalent to 5 half-lives (t1/2) of the agent (whichever is longer);
* Subjects who have or have undergone the following gastrointestinal disorders or procedures:
* Inflammatory bowel disease.
* Chronic faecal incontinence.
* History of chronic constipation or constipation in the 4 weeks prior to the screening phase (defined as 2 or less defaecations per week; associated with straining/passage of hard stools).
* Anal abscess.
* A history of radiation therapy to the pelvis.
* Fixed anal stenosis/fibrosis.
* Subjects with a history of neoplastic disease within 5 years (except for basal cell carcinoma or non-metastatic squamous cell carcinoma of the skin).
* Subjects with a clinically significant history of renal, hepatic, neurological, dermatological, immunological, major psychiatric (including drug or alcohol abusers), or haematological illness.
* Subjects with any laboratory tests considered clinically significant at screening.
* Subjects with planned elective or other treatment requiring hospitalisation, during the study, booked before entry into the study
* Subjects who will be unavailable for the duration of the trial, likely to be noncompliant with the protocol, or who are felt to be unsuitable by the Investigator for any other reason;
* Women of childbearing potential unless surgically sterile or using adequate contraception (IUD, oral or depot contraceptive, or barrier plus spermicide). Women using oral contraception must have started using it at least 2 months prior to enrolment.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Jordan, PhD, Study Director — S.L.A. Pharma
Locations (27):
- Bulgaria (6):
  - Dr Kantcho Kostadinov, Sevileva, Sevilieva
  - Vth MHAT, Sofia
  - MHAT Alexandrovska EAD, Sofia
  - Military Medical Academy, Sofia
  - D Rusev, Sofia
  - General Hospital for Active Treatment "Stefan Cherkezov", Veliko Tarnovo
- Germany (5):
  - Praxis, Blankenhain
  - Praxis, Fürth
  - End- und Dickdarm-Zentrum Mannheim, Mannheim
  - Gemeinschaftspraxis, Marl
  - Practice of Internal Medicine, Wiesbaden
- Lithuania (3):
  - Kaunas Medical University Clinics, Kaunas
  - Siauliai Hospital, Šiauliai
  - UAB Baltic and American Medical and Surgical Clinic, Vilnius
- Romania (10):
  - Spitalul Clinic de Urgenta "Prof Dr O Fodor" Cluj, Cluj Nopoca
  - Spitalul Clinic de Urgenta "Prof. Dr O Fodor", Cluj-Napoca
  - Spitalul Judetean de Urgenta Deva, Deva
  - Institutul de Gastroenterologie si Hepatologie lasi, Lasi
  - Spitalul Clinic Judetean de Urgente "Sf.Spiridon" lasi, Lasi
  - Cabinet Medical "Dr Lokos" Chirurgie Generala, Miercurea-Ciuc
  - Spitalul Clinic Judetean Mures, Tg Mures
  - Centrul Medical Tuculanu SRL, Timișoara
  - Spitalul Clinic Judetean de Urgenta Timisoara, Timișoara
  - Salvo-San-Ciobanca SRL, Zalău
- Hospital Clinico Universitario Lozano Blesa, Zaragoza, Spain
- United Kingdom (2):
  - Derby City General Hospital, Derby, Derbyshire
  - Royal Sussex County Hospital, Brighton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out-patient clinics
Pre-assignment Details: one week run-in period
Groups:
- Diltiazem Hydrochloride 2% Cream: 2.5 cm of Diltiazem hydrochloride 2% cream applied peri-anally three times daily for eight weeks.
  Diltiazem hydrochloride 2% cream : 3 times daily
- Diltiazem Hydrochloride 4% Cream: 2.5 cm Diltiazem hydrochloride 4% cream applied peri-anally three times daily for eight weeks.
  Diltiazem hydrochloride 4% cream : 3 times daily
- Placebo Cream: 2.5 cm placebo cream applied peri-anally three times daily for eight weeks.
  Placebo : 3 times daily
Period: Overall Study
Arm/Group | Diltiazem Hydrochloride 2% Cream | Diltiazem Hydrochloride 4% Cream | Placebo Cream
Started | 154 | 156 | 155
Completed | 147 | 148 | 145
Not Completed | 7 | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diltiazem Hydrochloride 2% Cream | Diltiazem Hydrochloride 4% Cream | Placebo Cream | Total
Number analyzed (Participants) | 154 | 156 | 155 | 465
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 145 | 146 | 149 | 440
  >=65 years | 9 | 10 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (14.2) | 42.5 (13.6) | 43.2 (12.5) | 43.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 96 | 87 | 263
  Male | 74 | 60 | 68 | 202
Region of Enrollment [Number; unit: participants]
  Spain | 3 | 2 | 4 | 9
  Romania | 101 | 105 | 103 | 309
  Lithuania | 5 | 6 | 6 | 17
  Bulgaria | 28 | 28 | 30 | 86
  Germany | 12 | 10 | 8 | 30
  United Kingdom | 5 | 5 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average of Worst Anal Pain Associated With or Following Defaecation for Week 4 (for the 7 Treatment Days Immediately Preceding the Week 4 Visit).
Description: Change from baseline in average of worst anal pain associated with or following defaecation for Week 4 (for the 7 treatment days immediately preceding the Week 4 visit). Numerical Rating Scale, range 0-10 where 0 = no pain and 10 = worst pain imaginable.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Diltiazem Hydrochloride 2% Cream | Diltiazem Hydrochloride 4% Cream | Placebo Cream
Number analyzed (Participants) | 154 | 156 | 155
units on a scale | -2.63 (0.15) | -2.64 (0.15) | -2.20 (0.15)

2. Secondary Outcome: Patient's Global Impression of Improvement (PGI-I)
Description: Compared to the way you felt prior to starting the study treatment, how would you now describe your problems related to the anal fissure?" Responses will be measured on a 7-point Likert scale where 1 = substantially worse, 2 = moderately worse, 3 = slightly worse, 4 = no change, 5 = slightly improved, 6 = moderately improved, and 7 = substantially improved. Percentage of subjects scoring 5,6 or 7 was assessed.
Time Frame: 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Diltiazem Hydrochloride 2% Cream | Diltiazem Hydrochloride 4% Cream | Placebo Cream
Number analyzed (Participants) | 154 | 156 | 155
percentage of participants | 62.4 | 51.9 | 46.5

3. Secondary Outcome: Assessment of Adverse Events, Clinical Laboratory Results, Vital Signs and Sensitivity Reactions
Description: Number of subjects with adverse events, abnormal clinical laboratory results, vital signs and occurrence of any local sensitivity reactions. Data are presented where the incidence is greater than or equal to 5%.
Time Frame: 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Diltiazem Hydrochloride 2% Cream | Diltiazem Hydrochloride 4% Cream | Placebo Cream
Number analyzed (Participants) | 154 | 156 | 155
percentage of participants | 70.1 | 70.5 | 60.6

ADVERSE EVENTS:
Time Frame: Throughout treatment period.
Description: Adverse events were recorded in the patient diary. For clarity adverse events recorded here are listed by organ system.
Arm/Group | Diltiazem Hydrochloride 2% Cream | Diltiazem Hydrochloride 4% Cream | Placebo Cream
Serious Adverse Events (participants affected / at risk) | 0/154 | 1/156 | 0/155
Other Adverse Events (participants affected / at risk) | 108/154 | 110/156 | 94/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diltiazem Hydrochloride 2% Cream (N=154) | Diltiazem Hydrochloride 4% Cream (N=156) | Placebo Cream (N=155)
Stapled haemorrhoidopexy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — post treatment prolapsed haemorrhoids required intervention.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diltiazem Hydrochloride 2% Cream (N=154) | Diltiazem Hydrochloride 4% Cream (N=156) | Placebo Cream (N=155)
Gastrointestinal disorders (Gastrointestinal disorders) | 91 (260) | 102 (296) | 84 (283)
Nervous system disorders (Nervous system disorders) | 20 (34) | 27 (40) | 23 (47)
Infections and infestations (Infections and infestations) | 11 (12) | 13 (20) | 6 (8)
General disorders and administration site conditions (General disorders) | 5 (6) | 6 (6) | 8 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less